CLINICAL TRIAL: NCT02408172
Title: The Study Was Approved by the Ethics Committee of Our Institution, Which is Accredited by the Office of Human Research Protection as an Institutional Review Board
Brief Title: Effects of Metoprolol and Amlodipine on Cardiac Remodeling, Arrhythmias and Blood Pressure Variation in Hypertensive Patients With Sleep Apnea Syndrome
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Harbin Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OSA-HT-1
Record Dates: First submitted 2015-03-12; First posted 2015-04-03 (Estimated); Last update posted 2017-02-15 (Actual); Status verified 2014-10

CONDITIONS: Sleep Apnea Syndrome; Hypertension
Keywords: hypertension; Sleep apnea syndrome; Amlodipine; metoprolol
MeSH Terms: conditions — Sleep Apnea Syndromes; Hypertension | interventions — Amlodipine; Metoprolol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- OSA-amlodipine (Experimental): To observe the effects of amlodipine (5mg) on blood pressure variation after 12 weeks of treatment
  Interventions: Drug: Amlodipine
- OSA-metoprolol (Experimental): To observe the effects of metoprolol (47.5mg) on blood pressure variation after 12 weeks of treatment
  Interventions: Drug: metoprolol

INTERVENTIONS:
Drug: Amlodipine — Amlodipine was given orally in a dose of 5mg/day to treat patients in the OSA-amlodipine group for 12 weeks.
  Arms: OSA-amlodipine
Drug: metoprolol — Metoprolol was given orally in a dose of 47.5mg/day to treat patients in the OSA-metoprolol group for 12 weeks.
  Arms: OSA-metoprolol

SUMMARY:
Obstructive sleep apnea (OSA) is a highly prevalent chronic sleep disorder that affects 3% to 7% in middle aged individuals and increases with age. OSA has been identified as the most common secondary cause associated with resistant hypertension. There is evidence that compared with older patients, the risk of hypertension in OSA patients may be particularly pronounced in younger adult ones (less than 50 years).

Traditionally, cardiovascular risk stratification in hypertensive patients was based on the average blood pressure (BP) measured in the clinic. Accumulated data has shown that target-organ damage is related not only to 24-h mean intra-arterial BP, but also to BP variability (BPV) in subjects with essential hypertension. Growing evidence demonstrated that BPV has considerable prognostic value for all-cause mortality and cardiovascular outcomes, independent of average BP. In addition, it has been found that hypoxia condition in pneumoconiosis patients was closely associated with exaggerated BPV in ambulatory BP. However, the selections of antihypertensive drugs remain yet not very clearly for hypertensive patients combined with OSA.

DETAILED DESCRIPTION:
Obstructive sleep apnea (OSA) is a highly prevalent chronic sleep disorder that affects 3% to 7% in middle aged individuals and increases with age. It is considered an important independent contributing factor for the development of hypertension, diabetes and heart rhythm disorders. The prevalence of arterial hypertension has been reported to reach 50% of patients with OSA. OSA has been identified as the most common secondary cause associated with resistant hypertension. There is evidence that compared with older patients, the risk of hypertension in OSA patients may be particularly pronounced in younger adult ones (less than 50 years).

Traditionally, cardiovascular risk stratification in hypertensive patients was based on the average blood pressure (BP) measured in the clinic. Accumulated data has shown that target-organ damage is related not only to 24-h mean intra-arterial BP, but also to BP variability (BPV) in subjects with essential hypertension. Growing evidence demonstrated that BPV has considerable prognostic value for all-cause mortality and cardiovascular outcomes, independent of average BP. In addition, it has been found that hypoxia condition in pneumoconiosis patients was closely associated with exaggerated BPV in ambulatory BP. However, the selections of antihypertensive drugs remain yet not very clearly for hypertensive patients combined with OSA.

ELIGIBILITY:
Inclusion Criteria:

* Men aged between 18 and 75 included years old, and
* Postmenopausal women who are no more than 75 years older.
* Patients with essential mild to moderate uncomplicated hypertension (DBP<110mmHg and SBP<180mmHg measured with a validated automatic device in sitting position) after initiation or intensification of appropriate healthy lifestyle modification,
* Without antihypertensive treatment in 2 weeks.

Exclusion Criteria:

* History of cerebrovascular disease: ischemic stroke, cerebral haemorrhage and TIA.
* History of cardiovascular disease:unstable angina, myocardial infarction, coronary revascularization and congestive heart failure.
* History of renal impairment.
* History of Type I diabetes mellitus or Type II diabetes uncontrolled.
* History of liver impairment.
* History of alcoholism or drug abuse.
* Known symptomatic orthostatic hypotension.
* Contra-indications to treatment with investigate products.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2013-10; Primary Completion 2017-06 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
24-hour Ambulatory Blood Pressure Monitoring | up to 3 years

SECONDARY OUTCOMES:
24-hour continuous ambulatory electrocardiography | up to 3 years
Ultrasonic echocardiography | up to 3 years

CONTACTS AND LOCATIONS:
Locations (2):
- Portable polysomnography, Suzhou, Jiangsu, China
- Twenty-four-hour ambulatory BP monitoring, Budapest, Budapest, Hungary